CLINICAL TRIAL: NCT03204136
Title: Tacrolimus Versus Methotrexate as Rescue Therapy for Refractory Inflammatory Bowel Disease: an Open-label, Retrospective Study
Brief Title: Tacrolimus Versus Methotrexate as Rescue Therapy for Refractory Inflammatory Bowel Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Key Laboratory of Gastroenterology and Hepatology, Ministry of Health, China (Other Government)
Responsible Party: Principal Investigator, Zhanghan Dai, attending physician, Key Laboratory of Gastroenterology and Hepatology, Ministry of Health, China
Other Study IDs: shrjibdc20170401
Record Dates: First submitted 2017-06-11; First posted 2017-06-29 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- tarcolimus: refractory inflammatory bowel disease patents who used tarcolimus to induce and maintain remission
- methotrexate: refractory inflammatory bowel disease patents who used methotrexate to induce and maintain remission

SUMMARY:
Mesalazine, steroid, immunosuppressants and biologic agents are main medical treatments in treating inflammatory bowel diseases. Yet some patients develop severe side effects or initial invalid to conventional therapies. Some studies have already showed that tarcolimus and methotrexate are both effective in inducing and maintaining disease remission. Here we conduct a retrospective study to compare the efficancy of tarcolimus and methotrexate in treating refractory inflammatory bowel diseases as rescue therapy.

ELIGIBILITY:
Inclusion Criteria:

* Tarcolimus or methotrexate was used in refractory inflammatory bowel disease patents

Exclusion Criteria:

* Pregnant woman

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inflammatory bowel disease patients who are refractory or intolerance to conventional therapy (including mesalazine, steroid, azathioprine and biological agents). Tarcolimus or methotrexate was used in these patients.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
disease activity assessment after one year treatment | one year
  Disease activity is assessed through blood test, radiology and clinical for both Crohn's disease and ulverative colitis. We evaluate clinical response based on Crohn's disease activity index (CDAI) for CD and Mayo score for UC at the end of one year observation.

SECONDARY OUTCOMES:
The number of participants require surgical intervention during treatment and the number of participants with treatment-related adverse events. | one year
  The number of participants require surgical intervention during treatment and the number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Zhihua Ran, MD, Principal Investigator — Division of Gastroenterology and Hepatology, Key Laboratory of Gastroenterology and Hepatology, Ministry of Health；Shanghai Inflammatory Bowel Disease Research Center；Renji Hospital, School of Medicine, Shanghai Jiao Tong University; Shanghai Institute of
Locations (1):
- Division of Gastroenterology and Hepatology, Key Laboratory of Gastroenterology and Hepatology, Ministry of Health；Shanghai Inflammatory Bowel Disease Research Center；Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China